CLINICAL TRIAL: NCT01591863
Title: A Phase 2A, Multi-Center, Open-Label, Uncontrolled Study to Determine the Safety, Tolerability, and Pharmacokinetics of Fidaxomicin Oral Suspension or Tablets in Pediatric Subjects With Clostridium Difficile-associated Diarrhea (CDAD)
Brief Title: Safety, Tolerability, and Pharmacokinetics of Fidaxomicin in Pediatric Subjects With Clostridium Difficile-associated Diarrhea (CDAD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Optimer Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5119-010; OPT-80-206 (Other: Optimerpharma Study Number)
Record Dates: First submitted 2012-04-27; First posted 2012-05-04 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Clostridium Difficile-associated Diarrhea
Keywords: Clostridium difficile-associated diarrhea; CDAD; Pediatric
MeSH Terms: interventions — Fidaxomicin; OPT 80

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fidaxomicin (Experimental)
  Interventions: Drug: fidaxomicin

INTERVENTIONS:
Drug: fidaxomicin — 6 months-5 years 11 months: oral suspension, 32 mg/kg/day with a maximum dose of 400 mg/day, divided into two doses, every 12 hours for 10 days.
  6 years-17 years 11 months: tablets, 200 mg every 12 hours for 10 days.
  Other Names: Dificid, Dificlir, OPT-80; PAR-101

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and pharmacokinetics of fidaxomicin in pediatric subjects with Clostridium difficile-associated diarrhea (CDAD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female 6 months to 17 years 11 months of age, inclusive;
* Female subjects of childbearing potential must use adequate contraception
* Diagnosed with CDAD

Exclusion Criteria:

* Concurrent use of oral vancomycin or metronidazole or any other effective treatments for CDAD
* Fulminant colitis
* History of inflammatory bowel disease
* Pregnant or breast-feeding
* Need for concurrent use of some P-glycoprotein inhibitors during therapy

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2012-06-15 (Actual); Primary Completion 2014-03-07 (Actual); Study Completion 2014-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] O'Gorman MA, Michaels MG, Kaplan SL, Otley A, Kociolek LK, Hoffenberg EJ, Kim KS, Nachman S, Pfefferkorn MD, Sentongo T, Sullivan JE, Sears P. Safety and Pharmacokinetic Study of Fidaxomicin in Children With Clostridium difficile-Associated Diarrhea: A Phase 2a Multicenter Clinical Trial. J Pediatric Infect Dis Soc. 2018 Aug 17;7(3):210-218. doi: 10.1093/jpids/pix037. PMID 28575523

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fidaxomicin
Started | 38
Completed | 24
Not Completed | 14
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — recurrence | 9
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fidaxomicin
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: months] | 99.4 (68.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events.
Description: Number of participants with adverse events, as categorized by MedDRA.
Time Frame: Enrollment through end of study (Day 38-41)
Population: Subjects receiving any amount of study drug
Measure: Number; unit: participants
Arm/Group | Fidaxomicin
Number analyzed (Participants) | 38
participants | 28

2. Primary Outcome: Investigate Concentrations of Fidaxomicin in Plasma Samples.
Description: 3-5 hour plasma levels of fidaxomicin (mean)
Time Frame: 3-5 hours after administration
Population: Treated subjects with evaluable plasma pharmacokinetic data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fidaxomicin
Number analyzed (Participants) | 36
ng/mL | 13.363 (15.472)

3. Primary Outcome: Investigate Concentrations of Fidaxomicin in Fecal Samples.
Description: End of therapy fecal levels of fidaxomicin (mean)
Time Frame: End of Therapy; Day 10-11
Population: Treated subjects with evaluable fecal data
Measure: Mean (Standard Deviation); unit: microgram/g
Arm/Group | Fidaxomicin
Number analyzed (Participants) | 30
microgram/g | 3227.93 (2668.08)

4. Secondary Outcome: Evaluate the Clinical Outcome by Assessment of Clinical Response.
Description: Positive clinical response defined as resolution of diarrhea
Time Frame: Day 10
Population: Treated subjects with positive toxin assay result within 24 hours of enrollment
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Fidaxomicin
Number analyzed (Participants) | 38
percentage of subjects | 92.1 [83.5 to 100]

5. Secondary Outcome: Evaluate the Clinical Outcome by Assessment of Sustained Clinical Response.
Description: Positive clinical response without recurrence through the follow-up period
Time Frame: 28 days post-treatment
Population: Treated subjects with positive toxin assay result within 24 hours of enrollment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fidaxomicin
Number analyzed (Participants) | 38
percentage of participants | 65.8 [50.7 to 80.9]

6. Primary Outcome: Investigate Concentrations of the Main Metabolite OP-1118 in Plasma Samples.
Description: 3-5 hour plasma levels of OP-1118 (mean)
Time Frame: 3-5 hours after administration
Population: Treated subjects with evaluable plasma pharmacokinetic data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fidaxomicin
Number analyzed (Participants) | 36
ng/mL | 60.016 (152.196)

7. Primary Outcome: Investigate Concentrations of the Main Metabolite OP-1118 in Fecal Samples.
Description: End of therapy fecal levels of OP-1118 (mean)
Time Frame: End of Therapy; Day 10-11
Population: Treated subjects with evaluable fecal data
Measure: Mean (Standard Deviation); unit: microgram/g
Arm/Group | Fidaxomicin
Number analyzed (Participants) | 30
microgram/g | 865.49 (614.15)

ADVERSE EVENTS:
Time Frame: From informed consent through 30 days after the last administration of study treatment.
Arm/Group | Fidaxomicin
Serious Adverse Events (participants affected / at risk) | 9/38
Other Adverse Events (participants affected / at risk) | 17/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fidaxomicin (N=38)
Clostridium difficilie colitis (Infections and infestations) | 3
febrile neutropenia (Blood and lymphatic system disorders) | 1
Hematemesis (Gastrointestinal disorders) | 1
vomiting (Gastrointestinal disorders) | 2
adenovirus infection (Infections and infestations) | 1
clostridial infection (Infections and infestations) | 1
septic shock (Infections and infestations) | 1
gastrostomy failure (Injury, poisoning and procedural complications) | 1
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fidaxomicin (N=38)
abdominal pain upper (Gastrointestinal disorders) | 3
constipation (Gastrointestinal disorders) | 2
diarrhea (Gastrointestinal disorders) | 2
nausea (Gastrointestinal disorders) | 2
oesophagitis (Gastrointestinal disorders) | 2
vomiting (Gastrointestinal disorders) | 3
chest pain (General disorders) | 2
pyrexia (General disorders) | 4
nasopharyngitis (Infections and infestations) | 2
dehydration (Metabolism and nutrition disorders) | 2
headache (Nervous system disorders) | 2
urticaria (Skin and subcutaneous tissue disorders) | 2
hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication or other public presentation of results from this study requires prior review and written approval of the Sponsor. Draft abstracts, manuscripts, and materials for presentation at scientific meetings should be provided to the Sponsor at least 30 working days prior to submission deadlines. Authorship of publications resulting from this study will be based on generally accepted criteria for major medical journals.